CLINICAL TRIAL: NCT05237817
Title: If Adrenal Incidentalomas Have the Influences to Occur and Progress in Patients With Stroke
Brief Title: Association Between Stroke and Adrenal Incidentalomas
Acronym: ABSAI
Status: Recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: yanh-stroke&adrenal
Record Dates: First submitted 2021-11-01; First posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2021-04

CONDITIONS: Stroke; Adrenal Incidentaloma
Keywords: Adrenal Incidentaloma; Autonomous cortisol secretion; Stroke
MeSH Terms: conditions — Stroke; Adrenal incidentaloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cerebral infarction Group: Patients with cerebral infarction, and enrolled in our emergency or clinical department.
- Intracerebral hemorrhage Group: Patients with intracerebral hemorrhage, and enrolled in our emergency or clinical department.
- Subarachnoid hemorrhage Group: Patients with subarachnoid hemorrhage, and enrolled in our emergency or clinical department.

SUMMARY:
Adrenal incidentalomas (AIs) are commonly encountered in transsection imaging which purpose not for suspected adrenal disease. However, part of AIs in patients is associated with Stroke. Stroke is a diseases which could cause of disability and death worldwide. In clinical practice, detailed information about the association between stroke and AIs is not available. In this study, the investigators aimed to investigate the risk for disability and death in the large group of stroke patients with AIs.

DETAILED DESCRIPTION:
Background:

Adrenal incidentalomas (AIs) are commonly encountered in transsection imaging which purpose not for suspected adrenal disease. However, part of AIs in patients is associated with Stroke . The investigators aimed to investigate the risk for disability and death in the large group of stroke patients with AIs.

Objective:

To measure the association between stroke and levels of autonomous cortisol secretion in patients with AIs.

Design:

Part 1, Retrospective cohort study.

From April 1, 2021, to September 30, 2021, cohort patients with stroke were recruited in this study. The investigators assess the standardised incidence rate of AIs in all patients. Meanwhile, detail information about stroke disease、patient and AIs characteristics were record.

Part 2, Prospective cohort study.

From Mar 1, 2022, to Feb 29, 2024, cohort patients with stroke plane to recruit in this study. All patient receive the plasma cortisol level after a 1-mg dexamethasone suppression test. The investigators assess the standardised incidence rate of AIs in all patients. Meanwhile, detail information about stroke disease、patient and AIs characteristics would be record.

ELIGIBILITY:
Inclusion Criteria:

* stroke disease , such as Cerebral infarction、Intracerebral hemorrhage and Subarachnoid hemorrhage.

Exclusion Criteria:

* presence of metastatic cancer;
* AIs smaller than 1 cm;
* nonadenoma lesions, such as myelolipomas,hemorrhages, and cysts;
* oral glucocorticoid treatment with more than single doses in the past 3 months;
* use of inhaled steroids or medication affecting dexamethasone metabolism;
* systemic estrogen treatment.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Stroke disease, and erolled in our emergency or clinical department.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of Adrenal incidentalomas | 5 years
  Assess the standardised incidence rate of AIs in all patients with stroke
Plasma cortisol level | 5 years
  Plasma cortisol level after a 1-mg dexamethasone suppression test

SECONDARY OUTCOMES:
Diameter of Adrenal incidentalomas | 5 years
  Maximal axial diameter of adrenal incidentalomas by computed tomography scan; Millimetre as a metric unit of length in this study

CONTACTS AND LOCATIONS:
Overall Officials: Tong W Ou, Dr., Study Director — Department of Urology, Xuanwu Hospital, Capital Medical University
Locations (1):
- Hao Yan, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided
un-decided if corporation for multi-centers study in the future.

REFERENCES:
- [Background] Kjellbom A, Lindgren O, Puvaneswaralingam S, Londahl M, Olsen H. Association Between Mortality and Levels of Autonomous Cortisol Secretion by Adrenal Incidentalomas : A Cohort Study. Ann Intern Med. 2021 Aug;174(8):1041-1049. doi: 10.7326/M20-7946. Epub 2021 May 25. PMID 34029490
- [Background] Ebbehoj A, Li D, Kaur RJ, Zhang C, Singh S, Li T, Atkinson E, Achenbach S, Khosla S, Arlt W, Young WF, Rocca WA, Bancos I. Epidemiology of adrenal tumours in Olmsted County, Minnesota, USA: a population-based cohort study. Lancet Diabetes Endocrinol. 2020 Nov;8(11):894-902. doi: 10.1016/S2213-8587(20)30314-4. PMID 33065059
- [Background] Fassnacht M, Arlt W, Bancos I, Dralle H, Newell-Price J, Sahdev A, Tabarin A, Terzolo M, Tsagarakis S, Dekkers OM. Management of adrenal incidentalomas: European Society of Endocrinology Clinical Practice Guideline in collaboration with the European Network for the Study of Adrenal Tumors. Eur J Endocrinol. 2016 Aug;175(2):G1-G34. doi: 10.1530/EJE-16-0467. PMID 27390021